CLINICAL TRIAL: NCT04213794
Title: A Prospective Study of Heated Intra-Peritoneal Chemotherapy (H.I.P.E.C.) With Doxorubicin and Cisplatin in Pediatric Patients With Pelvic and Abdominal Tumors. The TOAST IT Trial (Trial Of Adjuvant Surgical Treatment With Intraperitoneal Chemotherapy)
Brief Title: Heated Intra-peritoneal Chemotherapy With Doxorubicin and Cisplatin for Abdominal for Pelvic Tumors in Pediatric Patients
Acronym: TOASTIT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1947; NCI-2019-08650 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1947 (Other: Mayo Clinic in Rochester); 18-010108 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Malignant Abdominal Neoplasm; Malignant Pelvic Neoplasm; Recurrent Colon Carcinoma; Recurrent Desmoplastic Small Round Cell Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Gastric Carcinoma; Recurrent Liposarcoma; Recurrent Malignant Mesothelioma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Rectal Carcinoma; Recurrent Rhabdomyosarcoma; Recurrent Sarcoma; Refractory Colon Carcinoma; Refractory Desmoplastic Small Round Cell Tumor; Refractory Fallopian Tube Carcinoma; Refractory Gastric Carcinoma; Refractory Liposarcoma; Refractory Malignant Mesothelioma; Refractory Ovarian Carcinoma; Refractory Primary Peritoneal Carcinoma; Refractory Rectal Carcinoma; Refractory Rhabdomyosarcoma; Refractory Sarcoma; Resectable Liposarcoma; Resectable Malignant Mesothelioma; Resectable Sarcoma
MeSH Terms: conditions — Pelvic Neoplasms; Colonic Neoplasms; Desmoplastic Small Round Cell Tumor; Fallopian Tube Neoplasms; Stomach Neoplasms; Liposarcoma; Mesothelioma, Malignant; Ovarian Neoplasms; Rectal Neoplasms; Rhabdomyosarcoma; Sarcoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cytoreduction Surgical Procedures; Doxorubicin; Hyperthermic Intraperitoneal Chemotherapy; sodium thiosulfate; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cytoreduction, HIPEC) (Experimental): Patients undergo cytoreduction. Patients also undergo HIPEC over 60 minutes consisting of doxorubicin and cisplatin. Patients then receive sodium thiosulfate IV over 12 hours. Patients also undergo CT scan, MRI or PET/CT scan and blood sample collection throughout study.
  Interventions: Drug: Cisplatin; Procedure: Cytoreductive Surgery; Drug: Doxorubicin; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Sodium Thiosulfate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Cisplatin — Undergo HIPEC with doxorubicin and cisplatin
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Cytoreductive Surgery — Undergo cytoreduction
  Other Names: Cytoreduction
Drug: Doxorubicin — Undergo HIPEC with doxorubicin and cisplatin
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC with doxorubicin and cisplatin
  Other Names: HIPEC
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric Acid Disodium Salt
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computed Tomography (CT); CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging; NMRI; Structural MRI; sMRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This early phase I trial studies how well heated intra-peritoneal chemotherapy with doxorubicin and cisplatin work for the treatment of abdominal or pelvic tumors that can be removed by surgery (resectable), does not respond to treatment (refractory), or has come back (recurrent). Heated intra-peritoneal chemotherapy is a procedure performed in combination with abdominal surgery for cancer that has spread to the abdomen. It involves the infusion of a heated chemotherapy solution that circulates into the abdominal cavity. Chemotherapy drugs, such as doxorubicin and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Heating a chemotherapy solution and infusing it directly into the abdomen may kill more cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of heated intra-peritoneal chemotherapy (HIPEC) with doxorubicin (DOXO) and cisplatin (CDDP) after surgical resection of pediatric pelvic and abdominal tumors.

II. To assess morbidity, hospital length of stay and peri-operative mortality outcomes for pediatric patients with intraperitoneal sarcoma undergoing hyperthermic intraperitoneal chemotherapy.

SECONDARY OBJECTIVE:

I. To assess complications and adverse events of HIPEC. II. Evaluate disease recurrence patterns: locoregional versus distant. III. Evaluate disease progression defined by radio-graphically visible nodules greater than 1.5 cm.

OUTLINE:

Patients undergo cytoreduction. Patients also undergo HIPEC over 60 minutes consisting of doxorubicin and cisplatin. Patients then receive sodium thiosulfate intravenously (IV) over 12 hours.

After completion of the study treatment, patients are followed every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have resectable, primary refractory or recurrent intra-abdominal or pelvic tumors based on imaging studies with measurable disease (>= 1 cm in 2 perpendicular planes), or primary tumor with peritoneal implants in whom no known other curative treatment exists, and/or patients not on up-front clinical trial
* Evidence of macroscopic or microscopic intra-peritoneal seeding (separate from the primary tumor) identified at the time of exploratory surgery with or without primary tumor resection
* Peritoneal cancer index (PCI) =< 20 and surgeons deem high likelihood of complete residual tumor stage R0 (R0) resection
* No evidence of distant metastases at the time of enrollment
* Histologies to be considered include: rhabdomyosarcoma, liposarcoma, sarcoma (other), ovarian cancer, fallopian tube cancer, gastric cancer, colon cancer, rectal cancer, mesothelioma, and desmoplastic small-round-cell tumor
* Patients must be 1-25 years of age at the time of entry into the study
* Patients may be included in the study independent of the regimen of previous surgical, radiation, or chemotherapy treatments administered. Given the increased risk of entero-cutaneous fistulae observed in patients treated with HIPEC AFTER radiation therapy, patients will be assessed for risk by radiation oncology
* Karnofsky / Lansky performance score of >= 40 or Eastern Cooperative Oncology Group (ECOG) performance score of 3 or less
* Platelet count >= 50,000 (independent of transfusion) (performed no later than 14 days before surgery)
* Prothrombin and partial thromboplastin times =< 1.2 X normal (performed no later than 14 days before surgery)
* Total bilirubin =< 2 X normal (performed no later than 14 days before surgery)
* Serum glutamic-oxaloacetic transaminase (SGOT) =< 2 X normal (performed no later than 14 days before surgery)
* Serum glutamate pyruvate transaminase (SGPT) =< 2 X normal (performed no later than 14 days before surgery)
* Lactate dehydrogenase (LDH) =< 2 X normal (performed no later than 14 days before surgery)
* Alkaline phosphatase =< 2 X normal (performed no later than 14 days before surgery)
* Neutrophil count >= 750 (performed no later than 14 days before surgery)
* Patients must have adequate renal function defined as creatinine clearance (performed no later than 14 days before surgery) or radioisotope GFR (glomerular filtration rate) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender less than the following values:

  * 1 to < 2 years 0.6mg/dL for both males and females
  * 2 to < 6 years 0.8mg/dL for both males and females
  * 6 to <10 years 1.0mg/dL for both males and females
* A signed informed consent form (and assent form when appropriate) approved by the Mayo Clinic (Institutional Review Board [IRB]) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

* Females who are pregnant or breast-feeding during the study period will be excluded
* Distant metastatic disease not limited to peritoneum:

  * Solid organ metastases (liver, central nervous system, lung)
  * Known bone marrow involvement
* No critical cumulative dose of previous chemotherapy (total anthracycline dose not >= 435 mg / m^2)
* Prior HIPEC within 3 months
* Patients with an active infection requiring treatment or having an unexplained febrile illness (Tmax > 99.5 Fahrenheit [F]), patients with known immune deficiency disorder or known human immunodeficiency virus infection
* Patients must not have any systemic illness which precludes them from being an operative candidate as determined by anesthesia preoperative evaluation. This includes but is not limited to, sepsis, liver failure, renal failure, cardiovascular failure, pulmonary failure
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacitation

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of cytoreductive surgery (CRS) with heated intra-peritoneal chemotherapy (HIPEC) in this patient population | Up to 6 months
  To assess the feasibility of heated intra-peritoneal chemotherapy (HIPEC) with doxorubicin (DOXO) and cisplatin (CDDP) after surgical resection of pediatric pelvic and abdominal tumors.

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of diagnosis of cancer up, assessed to 5 years
  Will be estimated using the Kaplan-Meier method. Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging. Patient contact may be contacted by telephone.
Disease-free survival (DFS) | From the time of diagnosis of cancer up to 5 years
  Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging. Patient contact may be contacted by telephone.
Peritoneal-free recurrence | From the time of diagnosis of cancer up to 5 years
  Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging. Patient contact may be contacted by telephone.
Incidence of morbidity | 30, 60, and, 90 days post-HIPEC procedure
  Will be measured using the Clavien Dindo scale and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Incidence of mortality | 30 days post-HIPEC procedure
  Will be tracked using NCI CTCAE version 5.
Hospital length of stay | Up to 5 years
  Will be tracked using NCI CTCAE version 5.
Estimated blood loss (EBL) | Up to 5 years
Operative time | Up to 5 years
Progression free survival (PFS) | From the time protocol treatment is initiated, assessed up to 5 years
  The PFS is defined as the time between initiation of protocol treatment and the first occurrence of disease. It will be defined radiologically.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio C. Gargollo, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials